CLINICAL TRIAL: NCT00156091
Title: A Multicenter, Randomized, Double-Blind, Flexible-Dose, Long-Term Extension Trial of the Safety and Maintenance of Effect of Asenapine Using Olanzapine Positive Control in Subjects Who Complete Protocols 041021 or 041022.
Brief Title: Long-Term Efficacy and Safety of Asenapine Using Olanzapine as a Positive Control (41512)(COMPLETED)(P05784)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P05784; Hera;; 41512
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine; asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Olanzapine 20 mg QD
  Interventions: Drug: Olanzapine
- 2 (Experimental): Asenapine 5 or 10 mg BID
  Interventions: Drug: Asenapine
- 3 (Other): Double-Blind subjects randomized to only placebo medication for 6 weeks in the short-term 041021 or 041022 asenapine trials, were randomized (double-blind) Into the long-term 041512 asenapine extension trial and received asenapine 5 mg BID for Week 1. After Week 1, subjects received asenapine (either 5 mg BID or 10 mg BID) for the remainder of the 52 week trial.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Olanzapine — 5- 20 mg QD
  Arms: 1
Drug: Asenapine — 5 or 10 mg BID
  Arms: 2
Other: Placebo
  Arms: 3

SUMMARY:
Schizophrenia is a brain disease. The primary features of schizophrenia are characterized by Positive symptoms (symptoms that should not be there, inability to think clearly, to distinguish reality from fantasy i.e., hearing voices) and Negative symptoms (a reduction or absence of normal behaviors or emotions, i.e., unable to manage emotions, make decisions and relate to others). Other symptoms include reduced ability to recall and learn new information, difficulty with problem solving, or maintaining productive employment. The symptoms of schizophrenia may be due to an imbalance in chemicals in the brain, primarily dopamine and serotonin, which enables brain cells to communicate with each other.

The clinical development of asenapine, as described in the 2007 IDB appears to have antipsychotic activity with superior symptomatic control compared to placebo and an improved safety profile compared to currently available neuroleptics. Its fast dissolving formulation may further add to treatment compliance. While various titration schedules have been used in previous studies, dose increases at 5 mg BID up to 10 mg BID have been well tolerated. Therefore, further exploration in a larger group of subjects with acute exacerbation of schizophrenia using an asenapine flexible dosing design ( 5 or 10 mg BID) will mimic actual clinical practice in a long-term 52-week extension trial.

ELIGIBILITY:
Inclusion Criteria:

* Completed the short-term trial ( 041021 or 021022)
* Continued to meet all demographic and procedural inclusion criteria of the short-term trial upon entry into this long-term extension trial
* Sign a written informed consent for the 041512 trial.
* Demonstrated an acceptable degree of compliance with trial medication in the short-term trials in the opinion of the investigator

Exclusion Criteria:

* CGI-S score of greater or equal to 6 ( severely psychotic)
* Occurrence(s) of AE or other clinically significant findings that would prohibit their continuation
* Met any of exclusion criteria regarding medical/psychiatric status listed in the short-term trials ( 041021 or 041022)
* Met exclusion criteria for medication status in short-term trials except for antidepressants and mood stabilizers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2005-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To assess long-term safety including overall symptoms (AEs; SAEs); Vital signs; ISST; EPS; and maintenance of effect; for asenapine with haloperidol control. | Weeks 1;2; 4; 8; 12; 16; 24; 32; 40; 52 (Endpoint)
Quality of Life and Patient Functionality (QLS; Q-LES-Q and PETIT) | Weeks 16; 32; 52(Endpoint)

SECONDARY OUTCOMES:
Pregnancy tests; Lab tests | Weeks 8; 16; 32; 52 (Endpoint)
Physical exams | Week 12; 24; 52 (Endpoint)
Neurocognition and cognitive functioning | Weeks 24 and 52 (Endpoint)
Weight and abdominal girth | Weeks 4;8;12; 16; 24; 32;40;52(Endpoint)
ECGs | Weeks 2;4;8;24;52(Endpoint)
Depression (CDSS) | Weeks 12; 24; 52 (Endpoint)